CLINICAL TRIAL: NCT04189484
Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 2: PCSK9 Inhibitors - Alirocumab and Evolocumab
Brief Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: PCSK9 Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SCR-007
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subjects; Pharmacokinetics; Pharmacodynamics
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — evolocumab; alirocumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (evolocumab or alirocumab) or placebo
Who Masked: Participant, Investigator
Masking Description: The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
  Subjects and staff will be blinded to treatment assignment during confinement. The blind will be maintained through a randomization schedule held by the dispensing pharmacist. Subjects and staff will be informed of a subject's end of study day when discharged from confinement. Subjects and staff will not be informed of the specific treatment arm assignment. The clinical research nurse will administer the subcutaneous study drug in unit dose containers that are not transparent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Arm A: Evolocumab low dose (Experimental): Single dose of evolocumab 21 mg subcutaneous (SC)
  Interventions: Biological: Evolocumab
- Arm B: Evolocumab intermediate low dose (Experimental): Single dose of evolocumab 35 mg SC
  Interventions: Biological: Evolocumab
- Arm C: Evolocumab intermediate high dose (Experimental): Single dose of evolocumab 70 mg SC
  Interventions: Biological: Evolocumab
- Arm D: Evolocumab high dose (Experimental): Single dose of evolocumab 140 mg SC
  Interventions: Biological: Evolocumab
- Arm E: Alirocumab low dose (Experimental): Single dose of alirocumab 15 mg SC
  Interventions: Biological: Alirocumab
- Arm F: Alirocumab intermediate low dose (Experimental): Single dose of alirocumab 25 mg SC
  Interventions: Biological: Alirocumab
- Arm G: Alirocumab intermediate high dose (Experimental): Single dose of alirocumab 50 mg SC
  Interventions: Biological: Alirocumab
- Arm H: Alirocumab high dose (Experimental): Single dose of alirocumab 100 mg SC
  Interventions: Biological: Alirocumab
- Arm I: Placebo (Placebo Comparator): Single dose of placebo SC
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Evolocumab — Evolocumab 21 mg administered SC
  Arms: Arm A: Evolocumab low dose
Biological: Evolocumab — Evolocumab 35 mg administered SC
  Arms: Arm B: Evolocumab intermediate low dose
Biological: Evolocumab — Evolocumab 70 mg administered SC
  Arms: Arm C: Evolocumab intermediate high dose
Biological: Evolocumab — Evolocumab 140 mg administered SC
  Arms: Arm D: Evolocumab high dose
Biological: Alirocumab — Alirocumab 15 mg administered SC
  Arms: Arm E: Alirocumab low dose
Biological: Alirocumab — Alirocumab 25 mg administered SC
  Arms: Arm F: Alirocumab intermediate low dose
Biological: Alirocumab — Alirocumab 50 mg administered SC
  Arms: Arm G: Alirocumab intermediate high dose
Biological: Alirocumab — Alirocumab 100 mg administered SC
  Arms: Arm H: Alirocumab high dose
Biological: Placebo — Placebo administered SC
  Arms: Arm I: Placebo

SUMMARY:
This study is designed to assess pharmacokinetics and pharmacodynamics of evolocumab and alirocumab across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 72 healthy subjects assigned to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (evolocumab and alirocumab ) or placebo.

DETAILED DESCRIPTION:
This study is designed to assess pharmacokinetics and pharmacodynamics of evolocumab and alirocumab, two monoclonal antibodies that inhibit proprotein convertase subtilisin/kexin type 9 (PCSK9), across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 72 healthy subjects assigned to one of four dose groups (low, intermediate low, intermediate high, and high) of each drug (evolocumab or alirocumab) or placebo. Evolocumab doses are 21, 35, 70, and 140 mg. Reslizumab doses are 15, 25, 50, and 100 mg . Each arm will include 8 subjects (4 male and 4 female).

Subjects will be admitted for treatment on day -1 and receive a single dose of study drug or placebo on day 1. Depending on the treatment arm, subjects will remain in confinement for one week and continue follow-up through day 42, 56, or 84.

Blood samples (approximately 5 mL per sample) will be collected for determination of plasma concentrations for study drug. Additional blood samples will be collected for lipid analysis and determination of low-density lipoprotein cholesterol (LDL-C) and apolipoprotein B (apoB) (5 mL per sample; pharmacodynamic measure) and exploratory proteomics analyses (5 mL per sample).

Safety evaluations will include adverse event (AE) monitoring, vital sign measurements, and physical examinations. All AEs reported by the subject or observed by the investigator or clinical research unit (CRU) staff will be recorded. Any AE reported after the informed consent is signed and before study drug application will be recorded as medical history.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an institutional review board (IRB)-approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 55 years of age, inclusive, who has a body mass index of 18.5 to 32 kg/m2, inclusive, at Screening.
3. Subject has a LDL-C level >=100 and <=190 mg/dL inclusive, at Screening.
4. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
5. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day -1).
6. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the last application of study drug.
7. Male subjects must agree to practice 1 highly effective method of birth control (as determined by the investigator or designee) from at least 1 month before Check in (Day-1) until at least 1 month after the last application of study drug.
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures as to complete the study.

Exclusion Criteria:

1. Subject is taking cholesterol medication (e.g. statins).
2. Subject is anemic (i.e., with hematocrit or hemoglobin less than the lower limit of normal) or has any chronic condition(s) that may impact blood sample collection.
3. Subject has had previous exposure to the biologic evolocumab or alirocumab.
4. Subject has a history of asthma.
5. Subject has a history of anaphylaxis from environmental exposures such as peanuts or bee stings.
6. Subject has an allergic history that includes urticaria, angioedema or respiratory coughing or bronchospasm.
7. Subject has a history of severe local reactions or generalized erythema from skin allergen testing.
8. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug.
9. Subjects are currently participating in another clinical study of an investigational drug or are have been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
10. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
11. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 hours of dosing. Subjects must refrain from ingesting these throughout the study.
12. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study. This includes subjects with any underlying medical conditions that put subjects at higher risk for coronavirus disease of 2019 (COVID-19) complications; per current Center for Disease Control and Prevention (CDC) recommendations this includes:

    * People with chronic lung disease or moderate to severe asthma
    * People who have serious heart conditions
    * People who are immunocompromised
    * Many conditions can cause a person to be immunocompromised, including cancer treatment, smoking, bone marrow or organ transplantation, immune deficiencies, poorly controlled HIV, and prolonged use of corticosteroids and other immune weakening medications
    * People with severe obesity (BMI of 40 or higher)
    * People with diabetes
    * People with chronic kidney disease undergoing dialysis
    * People with liver disease
13. Subject has any signs or symptoms that are consistent with COVID-19. Per current CDC recommendations this includes subjects with the symptoms cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
14. Subject tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a molecular diagnostic test performed prior to admission.
15. Subject has known or suspected allergies or sensitivities to any study drug.
16. Subject has clinical laboratory test results (hematology, serum chemistry lipid panel and comprehensive metabolic panel) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
17. Subject has a positive test result at Screening for human immunodeficiency virus (HIV) 1 or 2 antibody, hepatitis C virus load, hepatitis C virus antibodies, or hepatitis B surface antigen.
18. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
19. Female subjects are pregnant or lactating before enrollment in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Nalepinski, MPAS, PA-C, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as a part of manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as any eventual publications.
Supporting Information: Study Protocol, SAP
Time Frame: April, 2022. Materials will be available indefinitely

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 7 | 7
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [34 to 41] | 37 [32 to 48] | 40 [36 to 43] | 33 [31 to 38] | 39 [34 to 47] | 31 [27 to 40] | 36 [30 to 52] | 40 [28 to 42] | 41 [35 to 50] | 36 [31 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 2 | 3 | 3 | 3 | 3 | 3 | 28
  Male | 5 | 4 | 4 | 6 | 5 | 5 | 5 | 5 | 5 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 1 | 0 | 1 | 1 | 1 | 4 | 3 | 15
  Not Hispanic or Latino | 8 | 4 | 7 | 8 | 7 | 7 | 7 | 4 | 5 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 2 | 5 | 2 | 4 | 5 | 2 | 2 | 2 | 28
  White | 4 | 6 | 3 | 6 | 4 | 2 | 6 | 5 | 5 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 72
Body weight [Median (Inter-Quartile Range); unit: kg] | 82 [75 to 86] | 67 [66 to 76] | 84 [76 to 86] | 88 [84 to 97] | 85 [80 to 102] | 79 [72 to 92] | 86 [81 to 90] | 78 [67 to 87] | 76 [71 to 84] | 83 [72 to 89]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.7 [24.7 to 28.6] | 27.0 [24.5 to 28.6] | 28.7 [26.7 to 30.2] | 29.5 [27.5 to 31.9] | 30.1 [29.5 to 30.7] | 27.9 [25.7 to 28.8] | 28.6 [27.0 to 30.6] | 25.8 [24.2 to 28.6] | 26.8 [23.8 to 29.8] | 28.3 [25.3 to 30.1]

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Area Under Effect Curve (AUEC) for LDL-C for Evolocumab and Alirocumab
Description: The values and variability of AUEC for LDL-C at low, intermediate-low, intermediate-high, and high doses of evolocumab and alirocumab. AUEC was calculated as the baseline-subtracted area under the LDL-C concentration-time curve expressed in units of mg/(dL*day). More negative AUEC values represent greater reductions in LDL-C exposure from baseline. The standard deviation is noted in parentheses. For each subject and dose, the maximum decrease from baseline LDL-C was determined using all sampled timepoints. AUEC values were log-transformed and an ANCOVA model was used to calculate geometric means and 90% confidence intervals for each treatment group.
Time Frame: Day -1 and 0h (pre-dose), 24h (post-dose); once on Day 2, 3, 4, 5, 7, 10, 14, 21, 28, 35, and 42 for all Arms. Additionally, once on Day 56 for Arms C, D, G, H, & I; and once on Day 70 and 84 for Arms D, H, & I.
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: mg/dL*day
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 7 | 7
mg/dL*day | -380 (228) | -754 (573) | -866 (658) | -1832 (806) | -580 (360) | -581 (319) | -668 (828) | -1902 (361) | -350 (881)

2. Primary Outcome: Maximum Change From Baseline for LDL-C for Evolocumab and Alirocumab
Description: The values and variability of maximum change from baseline for LDL-C at low, intermediate low, intermediate high, and high doses of evolocumab and alirocumab
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 7 | 7
mg/dL | -27.7 (11.8) | -45.1 (26.9) | -49.9 (26.2) | -70.1 (25.0) | -35.8 (16.3) | -40.6 (8.1) | -47.9 (18.8) | -54.6 (12.1) | -30.1 (18.7)

3. Secondary Outcome: Baseline-adjusted AUEC for Apolipoprotein B (ApoB) for Evolocumab and Alirocumab
Description: The values and variability of AUEC for ApoB at low, intermediate-low, intermediate-high, and high doses of evolocumab and alirocumab. AUEC was calculated as the baseline-subtracted area under the ApoB concentration-time curve expressed in units of mg/(dL*day). More negative AUEC values represent greater reductions in ApoB exposure from baseline. The standard deviation is noted in parentheses. For each subject and dose, the maximum decrease from baseline ApoB was determined using all sampled timepoints. AUEC values were log-transformed and an ANCOVA model was used to calculate geometric means and 90% confidence intervals for each treatment group.
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: mg/dL*day
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 7 | 7
mg/dL*day | -207 (313) | -482 (434) | -676 (453) | -1094 (952) | -469 (290) | -462 (231) | -128 (536) | -1087 (707) | -428 (560)

4. Secondary Outcome: Maximum Change From Baseline for apoB for Evolocumab and Alirocumab
Description: The values and variability of maximal difference at a single time-point for ApoB at low, intermediate low, intermediate high, and high doses of evolocumab and alirocumab
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 7 | 7
mg/dL | 24 (12) | 32 (17) | 36 (15) | 46 (16) | 23 (9) | 29 (6) | 28 (8) | 37 (7) | 17 (7)

5. Secondary Outcome: Maximum Concentration (Cmax) for Evolocumab and Alirocumab
Description: The values and variability of Cmax at low, intermediate low, intermediate high, and high doses of evolocumab and alirocumab
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8,12, 24, hours post-dose; once on Day 2, 3, 4, 5, 6, 7, 10, 14, 21, 28, 35, and 42 for all Arms. Additionally, once on Day 56 for Arms C, D, G, H, & I; and once on Day 70 and 84 for Arms D, H, & I.
Population: Analysis population includes all subjects who did not discontinue before the end of study with at least one pharmacokinetic (PK) sample above the lower limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose
Number analyzed (Participants) | 3 | 6 | 7 | 8 | 8 | 8 | 7 | 7
ug/mL | 0.7 (28) | 0.5 (62) | 2.0 (54) | 6.2 (36) | 0.8 (27) | 1.7 (73) | 2.9 (61) | 6.9 (41)

6. Secondary Outcome: Area Under the Curve (AUC) for Evolocumab and Alirocumab
Description: The values and variability of AUC at low, intermediate low, intermediate high, and high doses of evolocumab and alirocumab
Time Frame: as for outcome 5
Population: Analysis population includes all subjects who did not discontinue before the end of study with at least one PK sample above the lower limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL*day
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose
Number analyzed (Participants) | 3 | 6 | 7 | 8 | 8 | 8 | 7 | 7
mg/dL*day | 2.4 (67) | 0.8 (91) | 12.9 (71) | 65.7 (57) | 8.3 (55) | 17.1 (57) | 38.5 (92) | 107.9 (58)

7. Secondary Outcome: Dose-response Parameters (Slope) for LDL-C Area Under the Effect Curve Models for Evolocumab and Alirocumab
Description: Model parameter (slope) for LDL-C area under the effect curve model: Mean slope value calculated after combining data from low, intermediate low, intermediate high, and high doses of evolocumab or alirocumab with placebo data. The units of measure for slope are mg/dL•day / (mg dose).
Time Frame: as for outcome 1
Population: Analysis population for each group was limited to those subjects administered evolocumab or placebo (the evolocumab group) or administered alirocumab or placebo (alirocumab) who completed the study. Results from subjects administered placebo were used in all analyses. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 10000 repetitions.
Measure: Mean (95% Confidence Interval); unit: mg/dL•day / (mg dose)
Groups:
- Evolocumab: Area Under the Effect Curve Model for LDL-C: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all evolocumab and placebo arms.
- Alirocumab: Area Under the Effect Curve Model for LDL-C: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all alirocumab and placebo arms.
Arm/Group | Evolocumab: Area Under the Effect Curve Model for LDL-C | Alirocumab: Area Under the Effect Curve Model for LDL-C
Number analyzed (Participants) | 38 | 37
mg/dL•day / (mg dose) | -11 [-15 to -6] | -15 [-21 to -9]

8. Secondary Outcome: Pharmacodynamic Model Parameter, Maximum Effect (Emax), for LDL-C Maximum Change From Baseline Models With Evolocumab and Alirocumab
Description: Model parameter (Emax) for LDL-C maximum change from baseline curve models calculated after combining data from low, intermediate low, intermediate high, and high doses of evolocumab or alirocumab with placebo data.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Evolocumab: Maximum Change From Baseline Model for LDL-C: Model-based analysis using individual subject baseline-subtracted maximum change from baseline results from all evolocumab and placebo arms.
- Alirocumab: Maximum Change From Baseline Model for LDL-C: Model-based analysis using individual subject baseline-subtracted maximum change from baseline results from all alirocumab and placebo arms.
Arm/Group | Evolocumab: Maximum Change From Baseline Model for LDL-C | Alirocumab: Maximum Change From Baseline Model for LDL-C
Number analyzed (Participants) | 38 | 37
mg/dL | 84 [55 to 113] | 62 [50 to 75]

9. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for LDL-C Maximum Change From Baseline Models With Evolocumab and Alirocumab
Description: Model parameter (ED50) for LDL-C maximum change from baseline curve models calculated after combining data from low, intermediate low, intermediate high, and high doses of evolocumab or alirocumab with placebo data.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Evolocumab: Maximum Change From Baseline Model for LDL-C | Alirocumab: Maximum Change From Baseline Model for LDL-C
Number analyzed (Participants) | 38 | 37
mg | 32 [0 to 66] | 14 [5 to 23]

ADVERSE EVENTS:
Time Frame: 42 days for subjects in treatment groups A, B, E, and F; 56 days for subjects in treatment groups C and G; and 84 days for subjects in treatment groups D, H, and I
Arm/Group | Arm A: Evolocumab Low Dose | Arm B: Evolocumab Intermediate Low Dose | Arm C: Evolocumab Intermediate High Dose | Arm D: Evolocumab High Dose | Arm E: Alirocumab Low Dose | Arm F: Alirocumab Intermediate Low Dose | Arm G: Alirocumab Intermediate High Dose | Arm H: Alirocumab High Dose | Arm I: Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 1/8 | 5/8 | 3/8 | 4/8 | 3/8 | 1/8 | 5/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Evolocumab Low Dose (N=8) | Arm B: Evolocumab Intermediate Low Dose (N=8) | Arm C: Evolocumab Intermediate High Dose (N=8) | Arm D: Evolocumab High Dose (N=8) | Arm E: Alirocumab Low Dose (N=8) | Arm F: Alirocumab Intermediate Low Dose (N=8) | Arm G: Alirocumab Intermediate High Dose (N=8) | Arm H: Alirocumab High Dose (N=8) | Arm I: Placebo (N=8)
Corneal abrasion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sneezing excessive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04189484/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT04189484/SAP_002.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT04189484/ICF_000.pdf